CLINICAL TRIAL: NCT07008976
Title: A Randomized, Open-label, Parallel-controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of TQB2102 for Injection Versus Trastuzumab Emtansine for Injection in Patients With HER2-positive Advanced Breast Cancer
Brief Title: Clinical Trial of TQB2102 for Injection Versus Trastuzumab Emtansine for Injection in HER2-positive Advanced Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2102-III-02
Record Dates: First submitted 2025-05-30; First posted 2025-06-06 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2102 Injection (Experimental): The drug is administered by intravenous infusion, at a dose of 6mg/kg each time. It is given once every 3 weeks, and each 3-week period constitutes one treatment cycle.
  Interventions: Drug: TQB2102 Injection
- Trastuzumab Emtansine for Injection (Active Comparator): The drug is administered by intravenous infusion, at a dose of 3.6mg/kg each time. It is given once every 3 weeks, and each 3-week period constitutes one treatment cycle.
  Interventions: Drug: Trastuzumab Emtansine for Injection

INTERVENTIONS:
Drug: TQB2102 Injection — TQB2102 Injection is a Human Epidermal Growth Factor Receptor 2 (HER2) bispecific antibody-drug conjugate.
  Arms: TQB2102 Injection
Drug: Trastuzumab Emtansine for Injection — Trastuzumab Emtansine for Injection is HER2-targeting antibody-drug conjugate (ADC).
  Arms: Trastuzumab Emtansine for Injection

SUMMARY:
This study adopted a randomized, open-label, positive drug-controlled, multi-center trial design. The primary endpoint was PFS evaluated by the Independent Review Committee (IRC). Eligible subjects were randomly assigned in a 1:1 ratio to receive either TQB2102 for injection or trastuzumab emtansine for injection.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily participated in this study, signed the informed consent form, and had good compliance;
* Age: 18 - 75 years old (at the time of signing the informed consent form); Eastern Cooperative Oncology Group (ECOG )score ≤ 1; Expected survival period exceeds 3 months;
* HER2-positive, unresectable, locally advanced or metastatic invasive breast cancer confirmed by histopathological or cytological examination;
* According to the 2018 version of the American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP )HumanEpidermalGrowthFactorReceptor2 (HER2) testing guidelines, HER2 positive is defined as: immunohistochemical result of 3+ or Fluorescence In Situ Hybridization (FISH) dual probe positive;
* The hormone receptor (HR) status has been clearly determined:

  a) According to the 2020 version of the ASCO/CAP guidelines, HR positive includes ER positive and/or PR positive, that is, the proportion of tumor cells with positive staining among all tumor cells is ≥ 1%.
* Received anti-HER2 monoclonal antibody and taxane drugs during the recurrence/metastasis stage.
* Disease progression occurred during or after the most recent treatment or intolerance.
* At least 1 line of treatment has been received in the recurrence/metastasis stage.
* According to the Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 standard, at least one measurable lesion exists.

Exclusion Criteria:

* Excluded are patients with known spinal cord compression or active central nervous system metastases .
* Patients with only skin and/or intracranial lesions as target lesions.
* Patients with adverse reactions from previous treatments that have not recovered to a CTCAE v5.0 grade score of ≤1.
* Patients with poorly controlled blood pressure (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg).
* Patients with major cardiovascular diseases
* Patients with a history of interstitial lung disease/pneumonia (non-infectious type) requiring steroid intervention treatment, or currently having interstitial lung disease/pneumonia, or those with suspected interstitial lung disease/pneumonia indicated by screening period imaging and cannot be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The Progression-Free Survival (PFS) evaluated by Independent Review Committee (IRC) | Up 30 months
  The PFS evaluation of TQB2102 for injection compared with Trastuzumab Emtansine for injection in HER2-positive, unresectable locally advanced or metastatic breast cancer patients who had previously received anti-HER2 monoclonal antibodies and taxane drugs was assessed by the Independent Imaging Review Committee (IRC).

SECONDARY OUTCOMES:
The PFS evaluated by the researchers | Up 30 months
  The efficacy of injectable TQB2102 compared to injectable Trastuzumab Emtansine in evaluating the progression-free survival (PFS) in HER2-positive, unresectable locally advanced or metastatic breast cancer patients who had previously received anti-HER2 monoclonal antibodies and taxane drugs was assessed by the researchers.
The Overall Survival (OS) evaluated by the researchers | Up to 5 years
  The efficacy of injectable TQB2102 compared to injectable Trastuzumab Emtansine, as evaluated by the researchers, in HER2-positive, unresectable locally advanced or metastatic breast cancer patients who had previously received anti-HER2 monoclonal antibodies and taxane drugs.
The Duration of Response (DOR) evaluated by the researchers | Up to 5 years
  The efficacy of injectable TQB2102 compared to injectable Trastuzumab Emtansine as evaluated by the researchers in HER2-positive, unresectable locally advanced or metastatic breast cancer patients who had previously received anti-HER2 monoclonal antibodies and taxane drugs was studied.
The Partial Response (PR) evaluated by the researchers | Up to 5 years
  The efficacy of PR-assessed TQB2102 injection compared with Trastuzumab Emtansine injection in HER2-positive, unresectable locally advanced or metastatic breast cancer patients who had previously received anti-HER2 monoclonal antibodies and taxane drugs was evaluated by the researchers.
The Objective Response Rate (ORR)evaluated by the researchers | Up to 5 years
  The efficacy of injectable TQB2102 compared to injectable Trastuzumab Emtansine in evaluating the objective response rate (ORR) was assessed in HER2-positive, unresectable locally advanced or metastatic breast cancer patients who had previously received anti-HER2 monoclonal antibodies and taxane drugs.
The Clinical Benefit Rate (CBR) evaluated by the researchers | Up to 5 years
  The efficacy of CBR evaluated injection TQB2102 compared to injection Trastuzumab Emtansine in HER2-positive, unresectable locally advanced or metastatic breast cancer patients who had previously received anti-HER2 monoclonal antibodies and taxane drugs was assessed by the researchers.
The incidence and severity of adverse events | Sign the informed consent form, and until 28 days after the last medication administration / before starting a new anti-tumor treatment (which ever occurs first))
  The proportion of patients experiencing adverse events, and these adverse events are defined by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Antibody-drug conjugate (ADC) | Cycle 2, Cycle 4, Cycle 8, Cycle 16 (Each cycle is 3 weeks)
  Evaluate the population pharmacokinetic (PK) characteristics of TOB2102 for injection in patients with HER2-positive, unresectable, locally advanced or metastatic breast cancer who have previously received anti-HER2 monoclonal antibodies and taxane drugs.
Total antibodies | Cycle 2, Cycle 4, Cycle 8, Cycle 16 (Each cycle is 3 weeks)
  Evaluate the population pharmacokinetic (PK) characteristics of TOB2102 for injection in patients with HER2-positive, unresectable, locally advanced or metastatic breast cancer who have previously received anti-HER2 monoclonal antibodies and taxane drugs.
The small molecule toxin TO22723 | Cycle 2, Cycle 4, Cycle 8, Cycle 16 (Each cycle is 3 weeks)
  The blood concentration of the small molecule toxin TO22723 in TOB2102.
The incidence rate of Anti-Drug Antibody (ADA) | Cycle 1, Cycle 2, Cycle 4, Cycle 8, Cycle 16, 28 days (±7 days) after the last administration (Each cycle is 3 weeks)
  Evaluate the immunogenicity of injectable TQB2102 in conditions such as ADA incidence rate. Subjects with HER2-positive, unresectable, locally advanced or metastatic breast cancer who have previously received anti-HER2 monoclonal antibodies and taxane drugs.

CONTACTS AND LOCATIONS:
Locations (31):
- China (31):
  - The First Affiliated Hospital of Anhui Medical University, Bengbu, Anhui
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Shunyi Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Hospital Of Lanzhou University, Lanzhou, Gansu
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Affiliated Cancer Hospital Of Guangxi Medical University, Nanning, Guangxi
  - Cancer Hospital Of Guizhou Medical University, Guiyang, Guizhou
  - Hainan General Hospital, Haikou, Hainan
  - The Fourth Hospital Of Hebei Medical University, Shijiazhuang, Hebei
  - Affiliated Cancer Hospital Of Harbin Medical University, Harbin, Heilongjiang
  - Jiamusi Tuberculosis Hospital (Jiamusi Tumor Hospital), Jiamusi, Heilongjiang
  - Anyang Cancer Hospital, Anyang, Henan
  - The First Affiliated Hospital Of Henan University Of Science & Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Chifeng Municipal Hospital, Chifeng, Inner Mongolia
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital Of Dalian Medical University, Dalian, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Affiliated Hospital Of Jining Medical University, Jining, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Dazhopu Central Hospital, Dazhou, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Hangzhou Cancer Hospital, Hangzhou, Zhejiang